CLINICAL TRIAL: NCT02306590
Title: Efficacy, Safety and Tolerability of High Lipid and Calorie Supplementation in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., Departement of Neurology, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIPCAL-ALS
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; survival time; ALS Functional Rating Scale; quality of life; survival
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Intervention (Experimental): High caloric fatty diet for drinking (100% lipids, 4.5 kcal/ml) 405 kcal/90 ml/day in addition to daily food intake and standard of care; corresponding to an additional intake of 45 g fat per day
  Interventions: Dietary Supplement: Calogen
- Placebo (Placebo Comparator): Placebo drinking solution 8 kcal/90ml/day in addition to daily food intake and standard of care
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Calogen
  Arms: Study Intervention
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the trial is to investigate the survival time (the time from randomization until death or date of end of the study) compared between control group and experimental group.

This is a prospective, multicenter, randomized, stratified, parallel-group, double-blind trial comparing placebo with high caloric fatty diet for drinking as add-on therapy to 100 mg riluzole in amyotrophic lateral sclerosis (ALS) in 200 enrolled patients. For entry, the El Escorial Criteria for the diagnosis of ALS will be used. The patients have to be stable on riluzole at least 4 weeks prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Possible, probable (clinically or laboratory supported) or definite ALS according to the revised version of the El Escorial criteria (Brooks et al. 2000)
* Disease duration < 36 months
* Vital capacity of more than 50% of normal (defined as slow vital capacity, best of three measurements)
* Age ≥18 years
* Continuously treated with 100 mg riluzole daily for at least four weeks
* Capable of thoroughly understanding all information given and giving full informed consent according to GCP
* Willing to complete a diet questionnaire throughout participation in the study

Exclusion Criteria:

* Simultaneous participation in another interventional clinical study
* Previous participation in a drug clinical trial where last intake of the trial drug was within the last 12 weeks
* Known sensitivity or intolerance to rape oil or sunflower oil, or components thereof
* Tracheostomy
* Patients with gastrostomy
* Pregnancy or breastfeeding
* Any medical condition known to have an association with motor neuron dysfunction which might confound or obscure the diagnosis of ALS
* Presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment.
* Evidence of a major psychiatric disorder or clinically evident dementia precluding evaluation of symptoms.
* Liable to be not cooperative or comply with study requirements as assessed by the investigator, or unable to be reached in the case of emergency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Survival in ALS-patients with study intervention compared to placebo | 18 months

SECONDARY OUTCOMES:
Change of total ALS functional rating scale revised (ALSFRS-R) | 18 months
Change of individual quality of life (SEIQoL) | 18 months
Change of the slow vital capacity (sVC) | 18 months
Time to tracheostomy or death (combined) | 18 months
Change of Body Mass Index (BMI) | 18 months
Change of Appetite-Score, Council of Nutrition appetite questionnaire (CNAQ) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert C. Ludolph, MD, Prof., Principal Investigator — University Ulm
Locations (11):
- Germany (11):
  - Department of Neurology, University of Ulm, Ulm, Baden-Wurttemberg
  - Department of Neurology, University of Wuerzburg, Würzburg, Bavaria
  - Department of Neurology, Medical School Hannover, Hanover, Lower Saxony
  - Department of Neurology, University of Rostock, Rostock, Mecklenburg-Vorpommern
  - Department of Neurology, TU Dresden, Dresden, Saxony
  - Department of Neurology, University of Halle-Wittenberg, Halle, Saxony-Anhalt
  - Department of Neurology, University of Jena, Jena, Thuringia
  - Department of Neurology, Humboldt University, Berlin
  - Neurologische Universitätsklinik Bergmannsheil, Bochum
  - Department für Neurologie - Klinik für Schlafmedizin und Neuromuskuläre Erkrankungen Universitätsklinikum Münster, Münster
  - Department of Neurology, DKD HELIOS Klinik, Wiesbaden

REFERENCES:
- [Derived] Witzel S, Frauhammer F, Steinacker P, Devos D, Pradat PF, Meininger V, Halbgebauer S, Oeckl P, Schuster J, Anders S, Dorst J, Otto M, Ludolph AC. Neurofilament light and heterogeneity of disease progression in amyotrophic lateral sclerosis: development and validation of a prediction model to improve interventional trials. Transl Neurodegener. 2021 Aug 26;10(1):31. doi: 10.1186/s40035-021-00257-y. PMID 34433481